CLINICAL TRIAL: NCT05988580
Title: Evaluation of Postprandial Glycemia After Eating a Pasta Dish Made With Resistant Starch.
Brief Title: Postprandial Glycemia After Eating a Pasta Dish Made With Resistant Starch.
Acronym: ALISSEC2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ALISSEC 2.0
Record Dates: First submitted 2023-08-04; First posted 2023-08-14 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2023-07

CONDITIONS: Postprandial Glycemia; Resistant Starch
Keywords: Resistant starch; Postprandial glycemia; Postprandial insulinemia; Pasta
MeSH Terms: interventions — Resistant Starch

STUDY DESIGN:
Intervention Model Description: Randomised, double blind crossover intervention
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The products (experimental and placebo), will be produced by an external producer, who will retain the codes. None of the researchers involved in the study development or analyses will know the association until the end of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Subjects will consume a pasta dish with 20-22% of resistant starch
  Interventions: Other: Pasta dish with resistant starch; Other: Original version of pasta dish
- Control group (Placebo Comparator): Subjects will consume the original version of pasta dish
  Interventions: Other: Pasta dish with resistant starch; Other: Original version of pasta dish

INTERVENTIONS:
Other: Pasta dish with resistant starch — Pasta dish with 20-22% of resistant starch
Other: Original version of pasta dish — Original pasta dish, not reinforced with resistant starch

SUMMARY:
Resistant starch partially resists hydrolyzation by digestive enzymes in humans. Consequently, it is not absorbed in the small intestine and goes directly to the large intestine, where it is fermented by the intestinal microbiota, acting as a prebiotic and stimulating the growth of beneficial bacteria in the colon. In addition, the effect of resistant starch on postprandial glucose metabolism is studying. Thus, the present research on healthy subjects has been proposed.

The main objective is to assess the effect on postprandial glycemia of eating a pasta dish made with resistant starch versus its original version.

For this purpose, a randomized, double blind crossover study has been designed.

Target sample size is 18 subjects.

DETAILED DESCRIPTION:
The arms of the study are two:

* Experimental group (pasta dish made with resistant starch).
* Control group (original pasta dish).

Volunteers who wish to participate in the study will be interviewed by phone to verify that they meet the main inclusion criteria. Volunteers who meet the main inclusion criteria will be invited to an information and screening visit to resolve any doubts. Volunteers who agree to participate in the study will sign the informed consent and will be randomly assigned to one of the two arms of the study.

The two visits (clinical investigation days) of the study will take place with the volunteers in a fasting state of 4 hours and separated by at least 1 week washout period. The day before the visit, volunteers won't be able to drink alcohol, drink and eat excessively, and/or sleep few hours. Both visits will consist of eating a pasta dish in a maximum of 15 minutes. Blood samples will be taken before eating and during the 2.5 hours after (30, 60, 90, 120 and 150 minutes), in order to analyze the evolution of blood glucose and insulin levels.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-65 years.
* Body mass index: 18.5-29.9 kg/m2
* Volunteers who like and feel good with the ingredients of the dish.
* Good physical and psychological state.
* Volunteers undergoing pharmacological treatment will be maintained if the dose is stable for at least 3 months before the start of the study, excluding treatments that alter gastrointestinal function or glucose metabolism.
* Subjects must be able to understand and be willing to sign the informed consent, and must comply with all the procedures and requirements of the study.
* No weight variations considered relevant (+/- 3kg) in the last 3 months.

Exclusion Criteria:

* Subjects with relevant functional or structural abnormalities of the digestive system, such as malformations, angiodysplasias, active peptic ulcers, chronic inflammatory or malabsorption diseases, hiatal hernia, reflux, etc.
* Subjects who have undergone surgical interventions with permanent sequelae in the digestive system (for example, gastroduodenostomy).
* Subjects with a high alcohol intake, more than 14 units (women) and 20 units (men).
* Women who are breastfeeding or pregnant.
* Subjects with liver disease.
* Subjects with some type of cancer or undergoing treatment for it, or who have not had a period of at least 5 years since its eradication.
* Subjects with allergies to any component of the product under study or any other food that interferes and makes it difficult to monitor the study.
* Subjects who present some type of cognitive and/or psychic impairment.
* Subjects in whom poor collaboration is expected or who, in the opinion of the investigator, have difficulties in following the study procedures.
* Subjects who work the night shift.
* Subjects who follow some type of supplementation that interferes with the study.
* Subjects who are immersed in some treatment for weight loss.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Balanced in men and women
Enrollment: 18 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2023-10-27 (Actual); Study Completion 2023-11-15 (Actual)

PRIMARY OUTCOMES:
Baseline blood glucose | 0 min in the Clinical investigation day 1 and Clinical investigation day 2 (at least 7 days after the clinical investigation day 1)
  Blood glucose levels before start eating the pasta dish in each clinical investigation day will be analyzed by biochemical autoanalyzer and reported in mg/dL.
Postprandial blood glucose | 30, 60, 90, 120 and 150 min after start eating the pasta dish in the Clinical investigation day 1 and Clinical investigation day 2
  Blood glucose levels after start eating the pasta dish in each clinical investigation day will be analyzed by biochemical autoanalyzer and reported in mg/dL.
Glycemia Area Under the Curve | Baseline, 30, 60, 90, 120 and 150 minutes in the Clinical investigation day 1 and Clinical investigation day 2
  Postprandial glycemia levels after eating pasta dish in each clinical investigation day will be analyzed biochemical autoanalyzer and reported in mg/dL. Glycemia AUC will be calculated by the trapezoidal rule.

SECONDARY OUTCOMES:
Insulinemia Area Under the Curve | Baseline, 30, 60, 90, 120 and 150 minutes in Clinical investigation day 1 and Clinical investigation day 2
  Postprandial insulin levels after eating pasta dish in each clinical investigation day will be analyzed by ELISA and reported in mU/L. Insulinemia AUC will be calculated by the trapezoidal rule.
Baseline blood insulin | 0 min in the Clinical investigation day 1 and Clinical investigation day 2
  Blood insulin levels before start eating the pasta dish in each clinical investigation day will be analyzed by ELISA and reported in mU/L.
Postprandial blood insulin | 30, 60, 90, 120 and 150 min after start eating in the Clinical investigation day 1 and Clinical investigation day 2.
  Blood insulin levels after start eating the pasta dish in each clinical investigation day will be analyzed by ELISA and reported in mU/L.
Body weight | Clinical Investigation Day 1 (before eat the pasta dish) and Clinical Investigation Day 2 (before eat the pasta dish)
  Weight of participants will be measured by bioimpedance and reported in kg
Height | Clinical Investigation Day 1 (before eat the pasta dish) and Clinical Investigation Day 2 (before eat the pasta dish)
  Height of participants will be measured by stadiometer and reported in m.
Body mass index | Clinical Investigation Day 1 (before eat the pasta dish) and Clinical Investigation Day 2 (before eat the pasta dish)
  Body mass index will be calculated as follows: weight (kg)/ height (cm)2.
Acceptance of pasta dish | Clinical Investigation Day 1 (after eat the pasta dish) and Clinical Investigation Day 2 (after eat the pasta dish)
  Pasta dish acceptance will be analyzed by acceptance questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Fermín I Milagro Yoldi, PhD, Principal Investigator — University of Navarra; Idoia Ibero-Baraibar, PhD, Study Chair — University of Navarra; Carlos J González-Navarro, PhD, Study Chair — University of Navarra; Miguel López-Yoldi, PhD, Study Chair — University of Navarra; Salomé Pérez Diez, Study Chair — University of Navarra; Blanca Martínez de Morentin, Study Chair — University of Navarra; José I Riezu-Boj, PhD, Study Chair — University of Navarra
Locations (1):
- Centre for Nutrition Research, Pamplona, Navarre, Spain

IPD SHARING:
Plan to Share IPD: No